CLINICAL TRIAL: NCT02569918
Title: Natural Sensory Feedback for Phantom Limb Modulation and Therapy
Brief Title: Use of Hand Prosthesis With Surface Electrical Stimulation for Treatment of Phantom Limb Pain
Acronym: EPIONE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Wassim Raffoul (Other)
Collaborators: Aalborg University Hospital (Other); University of Freiburg (Other); Université Montpellier (Other); Lund University (Other); Indiana University School of Medicine (Other); Novosense AB (Industry); Mxm-Obelia (Industry); Ecole Polytechnique Fédérale de Lausanne (Other); Universitat Autonoma de Barcelona (Other); Catholic University of the Sacred Heart (Other); Aalborg University (Other)
Responsible Party: Sponsor-Investigator, Prof. Wassim Raffoul, Professor, University of Lausanne Hospitals
Organization: University of Lausanne Hospitals (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EPIONE-602547-4; 602547 (Other Grant/Funding Number: FP7-HEALTH-2013-INNOVATION)
Record Dates: First submitted 2015-10-06; First posted 2015-10-07 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Phantom Limb Pain
Keywords: Neuroplasticity; Sensory Feedback; Transcutaneous electrical stimulation; Robotic hand
MeSH Terms: conditions — Phantom Limb

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Surface electrical stimulation (Experimental): Operation of hand prosthesis with surface electrical sensory feedback
  Interventions: Device: Surface electrical stimulation

INTERVENTIONS:
Device: Surface electrical stimulation — Surface electrical stimulation using the following experimental devices. 1) The CE-approved HASOMED electrical isolated stimulator (Rehastim). 2) Two hand prosthesis: the robotic hand "Azzurra" (Prensilia, Italy) and the robotic hand "Multi-sensory Prosthetic Hand" (Wessling robotics, Germany) 3) The EPIONE Psychophysical Testing Platform software for stimulator control. Surface stimulation therapy is provided while providing visual guidance to the subject.

SUMMARY:
Phantom limb pain (PLP) is a frequent consequence of amputation, and it is notoriously difficult to treat. Amputation usually follows traumatic injuries or surgery following vascular diseases, diabetes, osteomyelitis or tumours in cases where the loss of the limb is required for the survival of the patient. The loss of a limb or other body parts is usually followed by the sensation that the lost body part is still present and can be felt. These phenomena are called, respectively, phantom awareness and phantom sensation. In 50-80% of amputees neuropathic pain develops in the lost limb also referred to as phantom limb pain (PLP). PLP can be related to a certain position or movement of the phantom limb, and might be elicited or worsened by a range of physical factors (e.g. changes in the weather or pressure on the residual limb) and psychological factors (e.g. emotional stress). It is well known that most treatments available for PLP today, such as pharmacological, surgical, anaesthetic, psychological and other, are ineffective.

Today it is believed that phantom limb pain may be related to changes in the cortex of the brain. There is evidence that these changes may be modulated - or even reversed - by providing sensory input to the stump or amputation zone. For example, cortical reorganization and alleviation of phantom limb pain has been observed in amputees following intense use of a hand prosthesis. However, there is no consistent knowledge on which type of peripheral sensory feedback may be effective in affecting the cortical plasticity or on how to best apply the sensory feedback.

The aim of the proposed research is to create natural, meaningful sensations through providing non-invasive sensory feedback (i.e. surface electrical stimulation) and the effectiveness to alleviate phantom limb pain and restore the cortical neuroplastic changes.

DETAILED DESCRIPTION:
Purpose of the experiment Up to 50-80 % of persons with amputations experience pain in the part of the body that is missing. This phenomenon is called phantom limb pain. It is not clear today why phantom limb pain occurs, and since the pain can be difficult to treat, it can affect the quality of life. Other scientific studies have shown, that the use of electrical stimulation applied through surface electrodes, can assist to decrease or alleviate the phantom limb pain. The aim of this study is to investigate if surface electrical stimulation for a period of 3 months can decrease or alleviate the phantom limb pain.

Methods Before the study begins, it will be necessary to test if the participant can tolerate the electrical stimulation and that the participant fulfill all criteria for participating in the study. During the study, different electrical stimulation sequences will be applied. The participant will be asked to fill out a series of questionnaires before, during and after the electrical stimulation, to describe how the electrical stimulation is experienced, and if the stimulation had an effect on the phantom limb pain and phantom sensations. The participant will also be asked about their general mood to investigate if this has an effect on the pain. The brain signals of the participants will be measured twice with either surface electrodes or with a scanning technique, while the participant is thinking about moving the amputated arm/hand, while moving the healthy arm, or while receiving electrical stimulation.

Plan for the experiment The experiment will take place over a period of 3 months and consists of a series of measurement and intervention sessions planned in 2 phases (intensive and semi-intensive therapy). All sessions will take place at the University Hospital of Lausanne (CHUV), Switzerland.

Visit 0. Interview and meeting with the subject (before the experiment begins, 1 session, 1-2 hours). Before the experiment begins, the participant is invited to a meeting and interview with project responsible to inform the participant about the experiment.

Visit 1. Preliminary investigations (before the experiment starts, 1 session, maximum 3 hours pr session). Before the experiment starts, but after the participant has signed the informed consent, the investigators will test if the participant can tolerate the electrical stimulation.The evoked sensory feedback sensations over the hand, will be characterized by non-invasive, transcutaneous electrical stimulation of the peripheral nerves in different locations on the upper limb, both when stimulating single channel per at time, or several channels simultaneously. This session will allow to identify the electrical stimulation optimal parameters (amplitude, frequency and pulse-width) to induce sensations on the hand and how to modulate these sensations, close to natural pattern. A protocol to be integrated in a close-loop (bidirectional control) system of artificial hand will be developed. If all criteria for participation are fulfilled, the participation of the subject will be decided.

Week 1 to week 12. Experiments with the superficial stimulation and hand prosthesis control (sEH) will then be performed three days per week for up to 3 hours per day according to the daily experiment aims and the compliance of the subject. The duration of the experiments will be 3 months. sEH will be divided in two different phases:

1. intensive (from 1st to 6th week) ; during this period the experiments will be carried out three days per week;
2. semi-intensive (from 7th to 12th week); during this period the experiments will be carried out one to two consecutive days per week;

The stimulation protocol will be composed of different programs (Exp):

The program 1 (Exp1) of the experiment will be performed in order to characterize the best positions and parameters for the stimulation. The subjects will provide his/her feedback by means of a dedicated psychophysical platform specially designed for this purpose.

The program 2 (Exp2) will be performed with the aim of trying different combination of channels and to identify the best pattern to deliver the most natural and useful sensation.

After each stimulus is delivered with the different combination of electrodes, the participant will provide his/her feedback on the type, strength and location of the sensation (if any) through the psychophysical testing platform.

sEH programs (Exp 3) The investigators will test the possibility to drive the stimulation produced by electrical stimulator with the transformed signals from sensors in (or over) the robotic hand, which is voluntary controlled by the user.

If everything works, the investigators will then proceed with the therapeutic use of the robotic hand prosthesis. More specifically, they will ask the participant to perform several tasks (depending on capacity, availability and motivation):

i) execution of different force levels ii) Identification of objects physical properties iii) Embodiment tests (ownership) iv) Functional improvement tests (activities of daily living):

Risks, side effects and disadvantages Surface stimulation may cause muscle-contractions. Attachment of the surface electrodes may cause the skin to become red or irritated for some hours following the experiment. The type of electrical stimulation used in this experiment is not associated with any known risks or side effects. When the sensory threshold is determined (i.e., the lowest strength of the electrical stimulation that the participant can feel), it may feel unpleasant or painful for a short period of time, but the unpleasantness or pain will disappear as soon as the electrical stimulation stops. The electrical stimulation applied during the intervention period will be adjusted such that is it not painful.

Measurement of the brain signals using the functional magnetic resonance imaging technique (fMRI) is safe, and there are no known risks or side effects of this procedure. The participant may, however, find that being placed inside the scanner is unpleasant. Measurement of the brain signals with surface electrodes is also considered safe, and there are no known risks or side effects of this procedure. There may be risks associated with the experiment that are unknown to the investigators. Therefore, the participant are asked to inform the investigators if the participant experiences any health problems during the experiment. If any side effects are discovered by the investigators, the participant will be informed immediately.

Benefits of the experiment There will be no benefits for the subject by participation in the study. However, the participant may find that his/her phantom limb pain is alleviated during the experiment as a result of the electrical stimulation. However, it is not possible for the investigators to predict if the electrical stimulation will affect the phantom limb pain, when the effect will start, how large the effect will be, or how long the effect will last. It is not possible to offer the participants a permanent or lasting solution after termination of the study.

Exclusion from and suspension of the experiment If the participant, according to the assessment of the investigator, react unexpectedly on the procedures or in any other way are not suitable for continuing in the experiment, the participation in the experiment can be terminated at any time. In general, the experiment will be terminated if it turns out that the subjects in general cannot tolerate the procedures of the project or find the experiment too exhausting.

ELIGIBILITY:
Inclusion Criteria:

* Amputation or peripheral nerve damage of an upper limb.
* Injury should be in the chronic, stable phase, such that any traumatic injuries or surgical wounds have healed and the person apart from eventual phantom pain (PLP) is healthy and able to carry out experiment.
* Other treatments for PLP tried with poor results.
* Patient accepts the study protocol as explained by the physician.
* The subject experienced intractable PLP (i.e. pain in the denervated or missing extremity) of more than 6 on numerical rating scale (NRS) or visual analog scale (VAS) (0-10 scale). The frequency of PLP episodes presents more than once a week.
* Amputee subjects without PLP are eligible for part of the study that targets the sensory feedback induction within advanced bidirectional prosthesis control.

Exclusion Criteria:

* Cognitive impairment
* Current or prior psychological impairments: Major personality disturbance (i.e. borderline, antisocial), Major depression, Bipolar I.
* Pregnancy
* History of or active substance abuse disorder
* Acquired brain injury with residual impairment
* Intellectual Disability (IQ < 70)
* Prior neurological or musculoskeletal disease
* Current or prior dermatological conditions
* Excessive sensitivity to electrical stimulation with surface electrodes. People afraid of electrical stimulation or pain.
* People with other diseases which may affect the function of the nervous system. (Diabetes, HIV, Renal Failure)
* Patients implanted with pacemakers

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-02; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Phantom limb pain | Change in phantom limb pain perception between baseline measurements and 3 months
  The pain intensity will be assessed using visual analog scale (VAS)
Cortical reorganization | Change in cortical reorganization between baseline measurements and 3 months
  The cortical response to peripheral stimulation will be tracked using MRI

SECONDARY OUTCOMES:
Phantom limb pain | Change in neuropathic pain symptoms between baseline measurements and 3 months
  The pain symptoms wil be assessed using the neuropathic pain symptom inventory (NPSI)
Cortical reorganization | Change in in cortical reorganization between baseline measurements and 3 months
  The cortical response to peripheral stimulation will be tracked using EEG

CONTACTS AND LOCATIONS:
Overall Officials: Wassim Raffoul, Professor, Principal Investigator — University of Lausanne Hospitals
Locations (1):
- University of Lausanne Hospital CHUV, Lausanne, Canton of Vaud, Switzerland